CLINICAL TRIAL: NCT01291056
Title: Differential Effects of Clomiphene Citrate in Women Undergoing Superovulation: A Double-blind, Placebo-controlled, Crossover Study
Brief Title: Differential Effects of Clomiphene Citrate in Women Undergoing Superovulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jessica Pittman, M.D., University of Utah
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 00038807
Record Dates: First submitted 2010-11-09; First posted 2011-02-07 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Mood
Keywords: Clomiphene citrate; Mood symptoms; Infertility; Superovulation; Effects of clomiphene on mood
MeSH Terms: conditions — Infertility | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomphine (Active Comparator): Each participant will take assigned medication (clomiphene citrate 50mg or placebo) on days 3-7 of her menstrual cycle.
  Interventions: Drug: Clomiphene
- Placebo (Placebo Comparator): Each participant will take assigned medication (clomiphene citrate 50mg or placebo) on days 3-7 of her menstrual cycle.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Each participant will take assigned medication (clomiphene citrate 50mg or placebo) on days 3-7 of her menstrual cycle.
  Arms: Placebo
Drug: Clomiphene — Each participant will take assigned medication (clomiphene citrate 50mg or placebo) on days 3-7 of her menstrual cycle.
  Arms: Clomphine

SUMMARY:
Clomiphene citrate is commonly used for ovulation induction in women with anovulation, correction of luteal phase deficiency or for superovulation as empiric therapy for unexplained infertility. Superovulation using clomiphene, usually with intrauterine insemination, is usually regarded as first line therapy for unexplained infertility, infertility due to mild endometriosis, or infertility with mild or moderate compromise of the male factor. The side effect profile reported by some women using clomiphene citrate is similar to symptoms of premenstrual dysphoric disorder (PMDD), including tension, irritability, depressed mood, affective lability, lack of energy, difficulty concentrating, and physical symptoms such as breast tenderness, bloating, headache joint and muscle pain. Few studies have been performed to examine the relationship between clomiphene citrate and mood symptoms; however, these studies have been limited by their small sample size, potential for recall bias and lack of randomization. Moreover, the experience of infertility is dysphoric in and of itself. Therefore, a rigorous evaluation of whether, when in the cycle, and how often clomiphene is associated with mood changes is needed. Such a study would add to the body of literature on this topic in three important ways: 1) use of prospective data collection to more accurately identify commonly reported symptoms, 2) characterize the timing of symptom occurrence relative to treatment cycle, and 3) provide information relevant to planning of future studies involving targeted treatment of clomiphene citrate induced symptoms. If clomiphene use is shown to affect mood, the results would point to an important avenue for psychopharmacologic insight into relationships between mood and sex steroids.

OBJECTIVES:

Specific Aim #1: To identify psychological and physical symptoms experienced by women taking clomiphene citrate for superovulation in a prospective, placebo controlled trial setting.

Specific Aim #2: To determine whether measures of the emotional and physical state prior to the administration of clomiphene, predict the occurrence of mood changes during the five days of clomiphene administration and in the late follicular and luteal phases of the cycle in which clomiphene was administered.

DETAILED DESCRIPTION:
The aim of this study is to identify psychological and physical symptoms experienced by women taking clomiphene citrate for superovulation in a prospective setting.

Clomiphene citrate is commonly used for ovulation induction in women with anovulation, correction of luteal phase deficiency or for superovulation as empiric therapy for unexplained infertility1. While clomiphene citrate is generally well tolerated, common side effects have been reported including vasomotor flushes, breast tenderness, pelvic discomfort, and mood swings. Visual changes, such as palenopsia are rarely reported2. The side effect profile reported by some women using clomiphene citrate is similar to symptoms of premenstrual dysphoric disorder (PMDD). Symptoms of PMDD include tension, irritability, depressed mood, affective lability, lack of energy, difficulty concentrating, and physical symptoms such as breast tenderness, bloating, headache joint and muscle pain. Several validated scales have been used to record symptom occurrences and to characterize the timing of symptom occurrence relative to the menstrual cycle3.

The psychological and mood side effects of clomiphene citrate in women undergoing infertility treatment have been studied to a limited degree. One study reported mood swings in 9 out of 14 women surveyed4. Another small study found a higher frequency of irritability, mood swings, feeling down and bloating in women undergoing fertility treatment who were taking clomiphene citrate compared to no medication.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating women, ages 25-40, with regular menstrual cycles 23-35 days in length who elect to treat unexplained infertility using clomiphene citrate for superovulation combined with intrauterine insemination will be eligible for participation in this study.
* Eligible participants will be identified by physicians at the Utah Center for Reproductive Medicine at the University of Utah and will be provided written informed consent before being randomized to treatment groups.
* Male partner's semen analysis must show a sperm density of at least 10 million per ml, and motility of 20% or greater and normal morphology using World Health Organization (WHO) criteria.

Exclusion Criteria:

* Women with a history of depression or anxiety disorder requiring hospitalization or treatment lasting more than six months and women who currently or have received treatment during the previous six months for anxiety, depression or other psychiatric disorders listed in the 4th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) will be excluded.
* Women who have previously received treatment with clomiphene citrate will also be excluded from the study.
* Women using tobacco or illicit drugs will be excluded from study participation.
* Because the measurement tool used to measure symptoms has been validated only in women who can read and speak English, women who cannot speak and read English will not be eligible to participate in the study.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Pittman, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were identified by physicians at the Utah Center for Reproductive Medicine at the University of Utah and provided written informed consent before being randomized to treatment groups.
Groups:
- Clomiphene Citrate, Then Placebo: Clomiphene Citrate 50 milligrams daily, then Placebo daily
- Placebo, Then Clomiphene Citrate: Placebo, then Clomiphene Citrate 50 milligrams daily
Period: Intervention One (Menstraution Day 3-7)
Arm/Group | Clomiphene Citrate, Then Placebo | Placebo, Then Clomiphene Citrate
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout
Arm/Group | Clomiphene Citrate, Then Placebo | Placebo, Then Clomiphene Citrate
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Intervention Two (Menstration Days 3-7)
Arm/Group | Clomiphene Citrate, Then Placebo | Placebo, Then Clomiphene Citrate
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clomiphene Citrate, Then Placebo | Placebo, Then Clomiphene Citrate | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Follicular Cycle Total Behavioral Score for Calendar of Premenstrual Experiences (COPE) Self Assessment
Description: To identify behavioral symptoms experienced by women taking clomiphene citrate versus placebo for superovulation in a prospective setting.
Time Frame: 1 year
Population: The scale incorporates physical, behavioral and mental symptoms. Each participant will rate the symptom(s) from zero to three based off severity. Symptoms with zero means that no symptoms are present. Symptoms with three means that the symptoms are severe. Range 0 -75 per cycle day.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Clomiphene Citrate: Clomiphene Citrate 50 milligrams daily
- Placebo: Placebo
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 3 [0 to 6] | 5 [1 to 18]

2. Primary Outcome: Follicular Cycle Total Physical Score for Calendar of Premenstrual Experiences (COPE) Self Assessment
Description: To identify physical symptoms experienced by women taking clomiphene citrate versus placebo for superovulation in a prospective setting.
Time Frame: 1 Year
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 10 [2.25 to 14] | 8 [5 to 26]

3. Primary Outcome: Luteal Cycle Total Behavioral Score for Calendar of Premenstrual Experiences (COPE) Self Assessment
Description: as for outcome 1
Time Frame: 1 year
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 5 [0 to 14.5] | 2 [0 to 13]

4. Primary Outcome: Luteal Cycle Total Physical Score for Calendar of Premenstrual Experiences (COPE) Self Assessment
Description: as for outcome 2
Time Frame: 1 year
Population: The scale incorporates physical, behavioral and mental symptoms. Each participant will rate the symptom(s) from zero to three based off severity. Symptoms with zero means that no symptoms are present. Symptoms with three means that the symptoms are severe. Physical symptoms were calculated to give the total score. Range 0 -75 per cycle day.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 9 [3.25 to 15] | 9 [0 to 28]

ADVERSE EVENTS:
Groups:
- Placebo, Then Clomiphene Citrate: Placebo daily, then Clomiphene Citrate 50 milligrams daily
Arm/Group | Clomiphene Citrate, Then Placebo | Placebo, Then Clomiphene Citrate
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes